CLINICAL TRIAL: NCT05997563
Title: Adjunctive Vaginal Progesterone (Micronized Progesterone Effervescent Vaginal Tablet) in Management of Preterm Labor: A Randomized Controlled Trial
Brief Title: Adjunctive Vaginal Progesterone in Management of Preterm Labor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Professor Vorapong Phupong, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 681/2023
Record Dates: First submitted 2023-08-08; First posted 2023-08-18 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micronized progesterone (Active Comparator)
  Interventions: Drug: Micronized progesterone
- Control (No Intervention)

INTERVENTIONS:
Drug: Micronized progesterone — Vaginal micronized progesterone effervescent once daily until delivery
  Arms: Micronized progesterone

SUMMARY:
This study evaluates the addition of vaginal micronized progesterone effervescent to standard treatment in the treatment of preterm labor. Half of participants will receive vaginal micronized progesterone effervescent and standard treatment, while the other half will receive only standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy with gestational age 24-33 weeks 6 days
* preterm labor
* received treatment with tocolysis and corticosteroids

Exclusion Criteria:

* conditions that need immediate delivery such as fetal distress, chorioamnionitis
* have medical complications such as heart disease, seizure
* fetal anomalies
* cervical dilatation more than 5 cm
* allergy to progesterone
* contraindication to progesterone
* contraindication to tocolytic use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
latency period | 13 weeks
  time from preterm labor to delivery

SECONDARY OUTCOMES:
gestational age at delivery | 13 weeks
  mean gestational age at delivery
preterm delivery less than 34 weeks | 10 weeks
  percentage of preterm delivery less than 34 weeks
preterm delivery less than 37 weeks | 13 weeks
  percentage of preterm delivery less than 37 weeks
neonatal complications | 13 weeks
  percentage of newborn with RDS, IVH, NEC, death
side effects | 13 weeks
  percentage of side effects such as headache, nausea/vomiting
compliance | 13 weeks
  percentage of complete drug use
good satisfaction | 13 weeks
  percentage of good satisfaction
good quality of life | 13 weeks
  percentage of good quality of life
Time to the recurrence of uterine contractions | 13 weeks
  mean time to the recurrence of uterine contractions

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University
Locations (1):
- Vorapong Phupong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 171: Management of Preterm Labor. Obstet Gynecol. 2016 Oct;128(4):e155-64. doi: 10.1097/AOG.0000000000001711. PMID 27661654
- [Background] Coomarasamy A, Williams H, Truchanowicz E, Seed PT, Small R, Quenby S, Gupta P, Dawood F, Koot YE, Atik RB, Bloemenkamp KW, Brady R, Briley A, Cavallaro R, Cheong YC, Chu J, Eapen A, Essex H, Ewies A, Hoek A, Kaaijk EM, Koks CA, Li TC, MacLean M, Mol BW, Moore J, Parrott S, Ross JA, Sharpe L, Stewart J, Trepel D, Vaithilingam N, Farquharson RG, Kilby MD, Khalaf Y, Goddijn M, Regan L, Rai R. PROMISE: first-trimester progesterone therapy in women with a history of unexplained recurrent miscarriages - a randomised, double-blind, placebo-controlled, international multicentre trial and economic evaluation. Health Technol Assess. 2016 May;20(41):1-92. doi: 10.3310/hta20410. PMID 27225013
- [Background] Facchinetti F, Vergani P, Di Tommaso M, Marozio L, Acaia B, Vicini R, Pignatti L, Locatelli A, Spitaleri M, Benedetto C, Zaina B, D'Amico R. Progestogens for Maintenance Tocolysis in Women With a Short Cervix: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jul;130(1):64-70. doi: 10.1097/AOG.0000000000002065. PMID 28594783
- [Background] Coomarasamy A, Devall AJ, Cheed V, Harb H, Middleton LJ, Gallos ID, Williams H, Eapen AK, Roberts T, Ogwulu CC, Goranitis I, Daniels JP, Ahmed A, Bender-Atik R, Bhatia K, Bottomley C, Brewin J, Choudhary M, Crosfill F, Deb S, Duncan WC, Ewer A, Hinshaw K, Holland T, Izzat F, Johns J, Kriedt K, Lumsden MA, Manda P, Norman JE, Nunes N, Overton CE, Quenby S, Rao S, Ross J, Shahid A, Underwood M, Vaithilingam N, Watkins L, Wykes C, Horne A, Jurkovic D. A Randomized Trial of Progesterone in Women with Bleeding in Early Pregnancy. N Engl J Med. 2019 May 9;380(19):1815-1824. doi: 10.1056/NEJMoa1813730. PMID 31067371
- [Background] Piette PCM. The pharmacodynamics and safety of progesterone. Best Pract Res Clin Obstet Gynaecol. 2020 Nov;69:13-29. doi: 10.1016/j.bpobgyn.2020.06.002. Epub 2020 Jun 25. PMID 32739288
- [Background] ACOG Practice Bulletin No.142: Cerclage for the management of cervical insufficiency. Obstet Gynecol. 2014 Feb;123(2 Pt 1):372-379. doi: 10.1097/01.AOG.0000443276.68274.cc. PMID 24451674
- [Background] Cicinelli E, De Ziegler D, Morgese S, Bulletti C, Luisi D, Schonauer LM. "First uterine pass effect" is observed when estradiol is placed in the upper but not lower third of the vagina. Fertil Steril. 2004 May;81(5):1414-6. doi: 10.1016/j.fertnstert.2003.12.016. PMID 15136116
- [Background] Simunic V, Tomic V, Tomic J, Nizic D. Comparative study of the efficacy and tolerability of two vaginal progesterone formulations, Crinone 8% gel and Utrogestan capsules, used for luteal support. Fertil Steril. 2007 Jan;87(1):83-7. doi: 10.1016/j.fertnstert.2006.05.067. Epub 2006 Nov 1. PMID 17081536
- [Background] Shiba R, Kinutani M, Okano S, Kawano R, Kikkawa Y. Efficacy of four vaginal progesterones for luteal phase support in frozen-thawed embryo transfer cycles: A randomized clinical trial. Reprod Med Biol. 2019 Sep 16;19(1):42-49. doi: 10.1002/rmb2.12300. eCollection 2020 Jan. PMID 31956284
- [Background] Schumacher M, Liere P, Ghoumari A. Progesterone and fetal-neonatal neuroprotection. Best Pract Res Clin Obstet Gynaecol. 2020 Nov;69:50-61. doi: 10.1016/j.bpobgyn.2020.09.001. Epub 2020 Sep 8. PMID 33039311
- [Result] Norman JE, Marlow N, Messow CM, Shennan A, Bennett PR, Thornton S, Robson SC, McConnachie A, Petrou S, Sebire NJ, Lavender T, Whyte S, Norrie J; OPPTIMUM study group. Vaginal progesterone prophylaxis for preterm birth (the OPPTIMUM study): a multicentre, randomised, double-blind trial. Lancet. 2016 May 21;387(10033):2106-2116. doi: 10.1016/S0140-6736(16)00350-0. Epub 2016 Feb 24. PMID 26921136
- [Result] Martinez de Tejada B, Karolinski A. Vaginal progesterone for maintenance tocolysis: a systematic review and metaanalysis of randomized trials. Am J Obstet Gynecol. 2015 Sep;213(3):438-9. doi: 10.1016/j.ajog.2015.05.037. Epub 2015 May 21. No abstract available. PMID 26003056
- [Result] Ashoush S, El-Kady O, Al-Hawwary G, Othman A. The value of oral micronized progesterone in the prevention of recurrent spontaneous preterm birth: a randomized controlled trial. Acta Obstet Gynecol Scand. 2017 Dec;96(12):1460-1466. doi: 10.1111/aogs.13236. Epub 2017 Oct 19. PMID 28949010
- [Result] Hyett J, Asadi N, Zare Khafri M, Vafaei H, Kasraeian M, Salehi A, Saadati N, Bazrafshan K. The use of vaginal progesterone as a maintenance therapy in women with arrested preterm labor: a double-blind placebo-randomized controlled trial. J Matern Fetal Neonatal Med. 2022 Mar;35(6):1134-1140. doi: 10.1080/14767058.2020.1743662. Epub 2020 Mar 26. PMID 32216490
- [Result] Palacio M, Ronzoni S, Sanchez-Ramos L, Murphy KE. Progestogens as Maintenance Treatment in Arrested Preterm Labor: A Systematic Review and Meta-analysis. Obstet Gynecol. 2016 Nov;128(5):989-1000. doi: 10.1097/AOG.0000000000001676. PMID 27741193